CLINICAL TRIAL: NCT07140796
Title: "A Crossover Study Investigating the Effects of Gluteus Medius-Focused Blood Flow Restriction Training With or Without Radial Shockwave Therapy on Q-Angle and Plantar Pressure in Adults With Genu Varum"
Brief Title: Effects of Hip Blood Flow Restriction and Shockwave Therapy on Q-Angle and Plantar Pressure in Adults With Genu Varum
Acronym: BFR-GVQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sungjin Park (Other)
Responsible Party: Sponsor-Investigator, Sungjin Park, Principal Investigator, Sahmyook University
Organization: Sahmyook University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYU 2025-06-031-001; Sahmyook University (Other Grant/Funding Number: SYU 2025-06-031-001)
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Genu Varum
Keywords: Genu varum; Blood Flow Restriction; BFR Training; Radial Shockwave Therapy; Q-angle; Plantar pressure
MeSH Terms: conditions — Genu Varum | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: This study uses a crossover design in which each participant receives two different interventions-gluteus medius-focused blood flow restriction (BFR) training alone and BFR training combined with radial extracorporeal shockwave therapy (rESWT)-in randomized order, with a washout period between the phases.
Masking Description: This study is open label because both the participants and investigators are aware of the intervention being administered. Due to the physical nature of the interventions (exercise and shockwave therapy), blinding was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR Only (Experimental): Participants in this group will undergo blood flow restriction (BFR) training alone. BFR training will be performed using a thigh cuff at a pressure estimated based on the participant's thigh circumference and blood pressure. Squats will be performed with 15% of body weight and hip internal rotation at 15 degrees, twice per week for 4 weeks.
  Interventions: Behavioral: Blood Flow Restriction Training; Device: Radial Extracorporeal Shockwave Therapy
- BFR + Shockwave (Experimental): Participants in this group will receive a combination of blood flow restriction (BFR) training and radial extracorporeal shockwave therapy (rESWT). BFR training will be conducted as in the other arm. Additionally, rESWT will be applied to the gluteus medius region before each exercise session, with 2000 pulses per session, twice per week for 4 weeks.
  Interventions: Behavioral: Blood Flow Restriction Training

INTERVENTIONS:
Behavioral: Blood Flow Restriction Training — Participants perform squats with 15% of their body weight under blood flow restriction using a thigh cuff. Hip internal rotation is set at 15 degrees. The training is conducted twice a week for 4 weeks. Cuff pressure is estimated using a predictive formula based on thigh circumference and systolic blood pressure.
Device: Radial Extracorporeal Shockwave Therapy — Radial extracorporeal shockwave therapy (rESWT) is applied to the gluteus medius region prior to each exercise session. The protocol includes 2000 pulses per session, applied twice per week for 4 weeks, using a radial shockwave device.
  Arms: BFR Only

SUMMARY:
This study aims to investigate the effects of gluteus medius-focused blood flow restriction (BFR) training, with or without the addition of radial shockwave therapy, on lower limb alignment in adults with genu varum. The study uses a crossover design and evaluates changes in Q-angle(Quadriceps-angle) and plantar pressure as primary outcomes. All interventions are non-invasive and supervised, and the goal is to identify effective therapeutic strategies to improve biomechanical alignment in individuals with bowed legs.

DETAILED DESCRIPTION:
This study investigates the effects of gluteus medius-focused blood flow restriction (BFR) training with or without radial extracorporeal shockwave therapy (rESWT) on lower limb alignment in adults with genu varum. Genu varum, commonly known as bow-leggedness, can lead to altered biomechanical patterns and increased stress on the medial knee joint. Strengthening the hip muscles, particularly the gluteus medius, may contribute to improved alignment and postural stability.

Participants will undergo two different intervention phases in a crossover design. Each phase includes a 4-week intervention period, with a 2-week washout in between. The primary outcome measures are Q-angle (quadriceps angle) and plantar pressure distribution, which will be assessed before and after each intervention phase using validated measurement tools.

This study aims to determine whether BFR training alone or combined with shockwave therapy provides greater improvement in lower limb alignment in individuals with genu varum. All interventions will be supervised, non-invasive, and conducted in a clinical setting under standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 20 and 40 years
* Diagnosed with genu varum (inter-knee distance ≥ 3 cm in standing position)
* No pain or surgery history in lower extremities within the last 6 months
* Able to walk independently without assistance
* Provide written informed consent

Exclusion Criteria:

* Neurological or musculoskeletal disorders affecting gait or posture
* Current use of medication affecting musculoskeletal or circulatory function
* Previous surgery on the spine, pelvis, or lower limbs
* Contraindications to shockwave therapy or BFR training (e.g., thromboembolic - disorders, deep vein thrombosis, cancer, etc.)
* Participation in other clinical trials within the past month

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Plantar pressure Distribution | Baseline and 4 Weeks Post-intervention
  Plantar pressure will be assessed using the TPScan system while participants walk barefoot over the pressure mat. The system will analyze peak pressure, pressure-time integral, and center of pressure trajectory in both feet. Data will be collected under two conditions (BFR alone vs. BFR + rESWT), and compared to evaluate the effects of the intervention.

SECONDARY OUTCOMES:
Quadriceps Angle (Q-angle) | At Baseline and 4 Weeks After Each Intervention Period
  Q-angle will be measured using a goniometer with participants in the supine position and legs extended. The angle is defined by the intersection between the line from the anterior superior iliac spine (ASIS) to the center of the patella, and the line from the patella to the tibial tuberosity. Data will be collected before and after each intervention to assess changes in lower limb alignment.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Su Rehabilitation Medicine Manual & Exercise Therapy Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
"IPD will not be shared because the data are limited to a small sample of clinical patients and involve privacy-sensitive health information."